CLINICAL TRIAL: NCT02482051
Title: Ultra Rapid Culture Independent Detection of High-Priority Carbapenem Resistant Enterobacteriaceae Directly From Blood
Status: Completed | Type: Observational
Sponsor: Denver Health and Hospital Authority (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Accelerate Diagnostics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 15-0082; 1R01AI116993 (NIH)
Record Dates: First submitted 2015-06-23; First posted 2015-06-25 (Estimated); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Bacteremia; Enterobacteriaceae Infections
Keywords: Carbapenem-resistant Enterobacteriaceae; Accelerate ID/AST
MeSH Terms: conditions — Bacteremia; Enterobacteriaceae Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to develop a new and very rapid diagnostic test for identifying a certain type of bacteria called Enterobacteriaceae in blood. Rapid identification of bacteria will assist in decreasing the use of antibiotics and help more patients survive bacterial infections of the blood.

DETAILED DESCRIPTION:
It is our overall goal to develop a new diagnostic technology that will facilitate antibacterial stewardship to reduce selective pressure and improve patient outcomes. The Institute of Medicine has identified antibiotic resistance as one of the key microbial threats to health in the United States and has prioritized decreasing inappropriate use of antimicrobials as the primary solution to address this threat. The emergence of carbapenem resistance among Enterobacteriaceae (CRE) in the United States represents a recent and severe byproduct of excessive antimicrobial use with a high mortality rate in bacteremia. A major barrier toward decreasing use of antimicrobials is lack of sensitive and accurate rapid diagnostic tests for identifying bacterial etiologies of infection.

ELIGIBILITY:
Inclusion Criteria:

* Laboratory confirmed gram negative bacilli blood culture

Exclusion Criteria:

* Pregnancy
* Prisoner

Ages: 7 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hospitalized patients with bacterial blood infections.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2015-07; Primary Completion 2022-01 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Bacteria identification | 3 hours
  Accuracy of bacteria identification by the Accelerate ID/AST system compared to conventional microbiological methods of gram negative bacilli.
Accuracy of carbapenem susceptibility testing | 3 hours
  Accuracy of carbapenem susceptibility testing by the Accelerate ID/AST system compared to conventional microbiological methods of gram negative bacilli.

CONTACTS AND LOCATIONS:
Overall Officials: Connie S Price, MD, Principal Investigator — Denver Health Medical Center
Locations (2):
- United States (2):
  - University of Colorado Hospital, Aurora, Colorado
  - Denver Health Medical Center, Denver, Colorado